CLINICAL TRIAL: NCT01116986
Title: Project 2: Identifying Optimal Smoking Cessation Intervention Components
Brief Title: Identifying Optimal Smoking Cessation Intervention Components (Cessation)
Acronym: Cessation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Dean Health System (Other); Mercy Health System (Network); Wake Forest University Health Sciences (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: H-2009-0204; 9P50CA143188 (NIH)
Record Dates: First submitted 2010-04-27; First posted 2010-05-05 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Smoking; Smoking Cessation; Nicotine Dependence
Keywords: Smoking; Smoking Cessation; Nicotine
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (32):
- 1, Patch, Gum, Prequit, Min In-Person, Min Phone, 8Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, Prequit Nicotine Gum, Counseling before quit attempt, Minimal In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt; Drug: Pre-Quit Nicotine Patch + Pre-Quit Nicotine Gum
- 2, Patch, Gum, Prequit, Min In-Person, Int Phone, 16Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, Prequit Nicotine Gum, Counseling before quit attempt, Minimal In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt; Drug: Pre-Quit Nicotine Patch + Pre-Quit Nicotine Gum
- 3, Patch, Gum, Prequit, Int In-Person, Min Phone, 16Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, Prequit Nicotine Gum, Counseling before quit attempt, Intensive In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt; Drug: Pre-Quit Nicotine Patch + Pre-Quit Nicotine Gum
- 4, Patch, Gum, Prequit, Int In-Person, Int Phone, 8Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, Prequit Nicotine Gum, Counseling before quit attempt, Intensive In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt; Drug: Pre-Quit Nicotine Patch + Pre-Quit Nicotine Gum
- 5, Patch, Gum, No Prequit, Min In-Person, Min Phone, 16Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, Prequit Nicotine Gum, No Counseling before quit attempt, Minimal In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt; Drug: Pre-Quit Nicotine Patch + Pre-Quit Nicotine Gum
- 6, Patch, Gum, No Prequit, Min In-Person, Int Phone, 8Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, Prequit Nicotine Gum, No Counseling before quit attempt, Minimal In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt; Drug: Pre-Quit Nicotine Patch + Pre-Quit Nicotine Gum
- 7, Patch, Gum, No Prequit, Int In-Person, Min Phone, 8Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, Prequit Nicotine Gum, No Counseling before quit attempt, Intensive In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt; Drug: Pre-Quit Nicotine Patch + Pre-Quit Nicotine Gum
- 8, Patch, Gum, No Prequit, Int In-Person, Int Phone, 16Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, Prequit Nicotine Gum, No Counseling before quit attempt, Intensive In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt; Drug: Pre-Quit Nicotine Patch + Pre-Quit Nicotine Gum
- 9, Patch, No Gum, Prequit, Min In-Person, Min Phone, 16Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, No Prequit Nicotine Gum, Counseling before quit attempt, Minimal In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt; Drug: Pre-Quit Nicotine Patch
- 10, Patch, No Gum, Prequit, Min In-Person, Int Phone, 8Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, No Prequit Nicotine Gum, Counseling before quit attempt, Minimal In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt; Drug: Pre-Quit Nicotine Patch
- 11, Patch, No Gum, Prequit, Int In-Person, Min Phone, 8Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, No Prequit Nicotine Gum, Counseling before quit attempt, Intensive In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt; Drug: Pre-Quit Nicotine Patch
- 12, Patch, No Gum, Prequit, Int In-Person, Int Phone, 16Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, No Prequit Nicotine Gum, Counseling before quit attempt, Intensive In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt; Drug: Pre-Quit Nicotine Patch
- 13, Patch, No Gum, No Prequit, Min In-Person, Min Phone, 8Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, No Prequit Nicotine Gum, No Counseling before quit attempt, Minimal In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt; Drug: Pre-Quit Nicotine Patch
- 14, Patch, No Gum, No Prequit, Min In-Person, Int Phone, 16Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, No Prequit Nicotine Gum, No Counseling before quit attempt, Minimal In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt; Drug: Pre-Quit Nicotine Patch
- 15, Patch, No Gum, No Prequit, Int In-Person, Min Phone, 16Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, No Prequit Nicotine Gum, No Counseling before quit attempt, Intensive In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt; Drug: Pre-Quit Nicotine Patch
- 16, Patch, No Gum, No Prequit, Int In-Person, Int Phone, 8Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? Prequit Nicotine Patch, No Prequit Nicotine Gum, No Counseling before quit attempt, Intensive In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt; Drug: Pre-Quit Nicotine Patch
- 17, No Patch, Gum, Prequit, Min In-Person, Min Phone, 16Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? No Prequit Nicotine Patch, Prequit Nicotine Gum, Counseling before quit attempt, Minimal In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt; Drug: Pre-Quit Nicotine Gum
- 18, No Patch, Gum, Prequit, Min In-Person, Int Phone, 8Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? No Prequit Nicotine Patch, Prequit Nicotine Gum, Counseling before quit attempt, Minimal In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt; Drug: Pre-Quit Nicotine Gum
- 19, No Patch, Gum, Prequit, Int In-Person, Min Phone, 8Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? No Prequit Nicotine Patch, Prequit Nicotine Gum, Counseling before quit attempt, Intensive In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt; Drug: Pre-Quit Nicotine Gum
- 20, No Patch, Gum, Prequit, Int In-Person, Int Phone, 16Wk (Experimental): How effective is the following Intervention? No Prequit Nicotine Patch, Prequit Nicotine Gum, Counseling before quit attempt, Intensive In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt; Drug: Pre-Quit Nicotine Gum
- 21, No Patch, Gum, No Prequit, Min In-Person, Min Phone, 8Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? No Prequit Nicotine Patch, Prequit Nicotine Gum, No Counseling before quit attempt, Minimal In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt; Drug: Pre-Quit Nicotine Gum
- 22, No Patch, Gum, No Prequit, Min In-Person, Int Phone, 16Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? No Prequit Nicotine Patch, Prequit Nicotine Gum, No Counseling before quit attempt, Minimal In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt; Drug: Pre-Quit Nicotine Gum
- 23, No Patch, Gum, No Prequit, Int In-Person, Min Phone, 16Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? No Prequit Nicotine Patch, Prequit Nicotine Gum, No Counseling before quit attempt, Intensive In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt; Drug: Pre-Quit Nicotine Gum
- 24, No Patch, Gum, No Prequit, Int In-Person, Int Phone, 8Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? No Prequit Nicotine Patch, Prequit Nicotine Gum, No Counseling before quit attempt, Intensive In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt; Drug: Pre-Quit Nicotine Gum
- 25, No Patch, No Gum, Prequit, Min In-Person, Min Phone, 8Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? No Prequit Nicotine Patch, No Prequit Nicotine Gum, Counseling before quit attempt, Minimal In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt
- 26, No Patch, No Gum, Prequit, Min In-Person, Int Phone, 16Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? No Prequit Nicotine Patch, No Prequit Nicotine Gum, Counseling before quit attempt, Minimal In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt
- 27, No Patch, No Gum, Prequit, Int In-Person, Min Phone, 16Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? No Prequit Nicotine Patch, No Prequit Nicotine Gum, Counseling before quit attempt, Intensive In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt
- 28, No Patch, No Gum, Prequit, Int In-Person, Int Phone, 8Wk (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? No Prequit Nicotine Patch, No Prequit Nicotine Gum, Counseling before quit attempt, Intensive In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Counseling before quit attempt; Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt
- 29, No Patch, No Gum, No Prequit, Min In-Person, Min Phone, 16 (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? No Prequit Nicotine Patch, No Prequit Nicotine Gum, No Counseling before quit attempt, Minimal In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt
- 30, No Patch, No Gum, No Prequit, Min In-Person, Int Phone, 8W (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? No Prequit Nicotine Patch, No Prequit Nicotine Gum, No Counseling before quit attempt, Minimal In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Minimal In-person counseling during quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt
- 31, No Patch, No Gum, No Prequit, Int In-Person, Min Phone, 8W (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? No Prequit Nicotine Patch, No Prequit Nicotine Gum, No Counseling before quit attempt, Intensive In-person counseling during quit attempt, Minimal Phone counseling during quit attempt, 8Wk Medication duration during quit attempt
  Interventions: Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Minimal phone counseling during the quit attempt; Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt
- 32, No Patch, No Gum, No Prequit, Int In-Person, Int Phone, 16 (Experimental): This arm of the project will address the following question:
  How effective is the following Intervention? No Prequit Nicotine Patch, No Prequit Nicotine Gum, No Counseling before quit attempt, Intensive In-person counseling during quit attempt, Intensive Phone counseling during quit attempt, 16Wk Medication duration during quit attempt
  Interventions: Behavioral: Intensive in-person counseling during the quit attempt; Behavioral: Intensive phone counseling during the quit attempt; Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt

INTERVENTIONS:
Behavioral: Counseling before quit attempt — Participants randomized to this condition will have 20-minute in-person counseling sessions 1 and 3 weeks before their target quit day and a 20-minute phone counseling session 2 weeks before their target quit day. In the in-person counseling session, the case manager will address issues such as smoking reduction, withdrawal coping, environmental restrictions on smoking, intra-treatment social support, autonomous motivation, and practice quit attempts. Participants will be asked to engage in two practice quit attempts. These attempts will each last 8 hours and will be assigned (in collaboration with the smoker) to occur on one weekend day and one weekday the second and third weeks after the quit day.
  Arms: 1, Patch, Gum, Prequit, Min In-Person, Min Phone, 8Wk; 10, Patch, No Gum, Prequit, Min In-Person, Int Phone, 8Wk; 11, Patch, No Gum, Prequit, Int In-Person, Min Phone, 8Wk; 12, Patch, No Gum, Prequit, Int In-Person, Int Phone, 16Wk; 17, No Patch, Gum, Prequit, Min In-Person, Min Phone, 16Wk; 18, No Patch, Gum, Prequit, Min In-Person, Int Phone, 8Wk; 19, No Patch, Gum, Prequit, Int In-Person, Min Phone, 8Wk; 2, Patch, Gum, Prequit, Min In-Person, Int Phone, 16Wk; 20, No Patch, Gum, Prequit, Int In-Person, Int Phone, 16Wk; 25, No Patch, No Gum, Prequit, Min In-Person, Min Phone, 8Wk; 26, No Patch, No Gum, Prequit, Min In-Person, Int Phone, 16Wk; 27, No Patch, No Gum, Prequit, Int In-Person, Min Phone, 16Wk; 28, No Patch, No Gum, Prequit, Int In-Person, Int Phone, 8Wk; 3, Patch, Gum, Prequit, Int In-Person, Min Phone, 16Wk; 4, Patch, Gum, Prequit, Int In-Person, Int Phone, 8Wk; 9, Patch, No Gum, Prequit, Min In-Person, Min Phone, 16Wk
Behavioral: Minimal In-person counseling during quit attempt — Participants randomized to minimal in-person counseling will receive one 3-minute in-person session occurring one week before their target quit day. The clinician will also inform the participant of the sort of phone counseling follow-up that s/he will receive in 1 and 2 weeks after their quit date. (This resembles the real-world situation in which the clinician discusses the sort of follow-up intervention a patient will receive.)
  Arms: 1, Patch, Gum, Prequit, Min In-Person, Min Phone, 8Wk; 10, Patch, No Gum, Prequit, Min In-Person, Int Phone, 8Wk; 13, Patch, No Gum, No Prequit, Min In-Person, Min Phone, 8Wk; 14, Patch, No Gum, No Prequit, Min In-Person, Int Phone, 16Wk; 17, No Patch, Gum, Prequit, Min In-Person, Min Phone, 16Wk; 18, No Patch, Gum, Prequit, Min In-Person, Int Phone, 8Wk; 2, Patch, Gum, Prequit, Min In-Person, Int Phone, 16Wk; 21, No Patch, Gum, No Prequit, Min In-Person, Min Phone, 8Wk; 22, No Patch, Gum, No Prequit, Min In-Person, Int Phone, 16Wk; 25, No Patch, No Gum, Prequit, Min In-Person, Min Phone, 8Wk; 26, No Patch, No Gum, Prequit, Min In-Person, Int Phone, 16Wk; 29, No Patch, No Gum, No Prequit, Min In-Person, Min Phone, 16; 30, No Patch, No Gum, No Prequit, Min In-Person, Int Phone, 8W; 5, Patch, Gum, No Prequit, Min In-Person, Min Phone, 16Wk; 6, Patch, Gum, No Prequit, Min In-Person, Int Phone, 8Wk; 9, Patch, No Gum, Prequit, Min In-Person, Min Phone, 16Wk
Behavioral: Intensive in-person counseling during the quit attempt — Participants randomized to intensive in-person counseling will receive three 20-minute face-to-face counseling sessions: one during the week before the target quit day, one on the target quit day and one during the week after the target quite day. The counseling will include intra-treatment social support and skill-based competence intervention components.
  Arms: 11, Patch, No Gum, Prequit, Int In-Person, Min Phone, 8Wk; 12, Patch, No Gum, Prequit, Int In-Person, Int Phone, 16Wk; 15, Patch, No Gum, No Prequit, Int In-Person, Min Phone, 16Wk; 16, Patch, No Gum, No Prequit, Int In-Person, Int Phone, 8Wk; 19, No Patch, Gum, Prequit, Int In-Person, Min Phone, 8Wk; 20, No Patch, Gum, Prequit, Int In-Person, Int Phone, 16Wk; 23, No Patch, Gum, No Prequit, Int In-Person, Min Phone, 16Wk; 24, No Patch, Gum, No Prequit, Int In-Person, Int Phone, 8Wk; 27, No Patch, No Gum, Prequit, Int In-Person, Min Phone, 16Wk; 28, No Patch, No Gum, Prequit, Int In-Person, Int Phone, 8Wk; 3, Patch, Gum, Prequit, Int In-Person, Min Phone, 16Wk; 31, No Patch, No Gum, No Prequit, Int In-Person, Min Phone, 8W; 32, No Patch, No Gum, No Prequit, Int In-Person, Int Phone, 16; 4, Patch, Gum, Prequit, Int In-Person, Int Phone, 8Wk; 7, Patch, Gum, No Prequit, Int In-Person, Min Phone, 8Wk; 8, Patch, Gum, No Prequit, Int In-Person, Int Phone, 16Wk
Behavioral: Minimal phone counseling during the quit attempt — Participants randomized to this condition will receive minimal phone counseling consisting of one 10-minute phone counseling session on the morning of the target quit day. This session will address motivation to quit, strategies for coping with urges to smoke and use of the medication, and will provide support. Thus, all participants will get some counseling support on the quit day, which reflects the fact that initial lapses often occur on the target quit day, and quit day smoking is an important determinant of ultimate outcome.
  Arms: 1, Patch, Gum, Prequit, Min In-Person, Min Phone, 8Wk; 11, Patch, No Gum, Prequit, Int In-Person, Min Phone, 8Wk; 13, Patch, No Gum, No Prequit, Min In-Person, Min Phone, 8Wk; 15, Patch, No Gum, No Prequit, Int In-Person, Min Phone, 16Wk; 17, No Patch, Gum, Prequit, Min In-Person, Min Phone, 16Wk; 19, No Patch, Gum, Prequit, Int In-Person, Min Phone, 8Wk; 21, No Patch, Gum, No Prequit, Min In-Person, Min Phone, 8Wk; 23, No Patch, Gum, No Prequit, Int In-Person, Min Phone, 16Wk; 25, No Patch, No Gum, Prequit, Min In-Person, Min Phone, 8Wk; 27, No Patch, No Gum, Prequit, Int In-Person, Min Phone, 16Wk; 29, No Patch, No Gum, No Prequit, Min In-Person, Min Phone, 16; 3, Patch, Gum, Prequit, Int In-Person, Min Phone, 16Wk; 31, No Patch, No Gum, No Prequit, Int In-Person, Min Phone, 8W; 5, Patch, Gum, No Prequit, Min In-Person, Min Phone, 16Wk; 7, Patch, Gum, No Prequit, Int In-Person, Min Phone, 8Wk; 9, Patch, No Gum, Prequit, Min In-Person, Min Phone, 16Wk
Behavioral: Intensive phone counseling during the quit attempt — Participants randomized to this condition will receive intensive phone counseling consisting of three 15-minute phone sessions (on the morning of the target quit day and on days 2 and 10 after the quit day). The content of the target quit day phone call will emphasize intra-treatment social support, skill execution and avoidance of danger situations. The quit day phone call is intended to augment any other clinician counseling received either on the phone or in person; such interventions tend to have additive effects and produce strong dose-response effects as a function of the duration of the counseling intervention.
  Arms: 10, Patch, No Gum, Prequit, Min In-Person, Int Phone, 8Wk; 12, Patch, No Gum, Prequit, Int In-Person, Int Phone, 16Wk; 14, Patch, No Gum, No Prequit, Min In-Person, Int Phone, 16Wk; 16, Patch, No Gum, No Prequit, Int In-Person, Int Phone, 8Wk; 18, No Patch, Gum, Prequit, Min In-Person, Int Phone, 8Wk; 2, Patch, Gum, Prequit, Min In-Person, Int Phone, 16Wk; 20, No Patch, Gum, Prequit, Int In-Person, Int Phone, 16Wk; 22, No Patch, Gum, No Prequit, Min In-Person, Int Phone, 16Wk; 24, No Patch, Gum, No Prequit, Int In-Person, Int Phone, 8Wk; 26, No Patch, No Gum, Prequit, Min In-Person, Int Phone, 16Wk; 28, No Patch, No Gum, Prequit, Int In-Person, Int Phone, 8Wk; 30, No Patch, No Gum, No Prequit, Min In-Person, Int Phone, 8W; 32, No Patch, No Gum, No Prequit, Int In-Person, Int Phone, 16; 4, Patch, Gum, Prequit, Int In-Person, Int Phone, 8Wk; 6, Patch, Gum, No Prequit, Min In-Person, Int Phone, 8Wk; 8, Patch, Gum, No Prequit, Int In-Person, Int Phone, 16Wk
Drug: Long Term Nicotine Patch+ Nicotine Gum During Quit Attempt — If randomized to this condition:
  After the target quit day:
  Patch:
  IF > 10 cigs/day: one 21 mg nicotine patch per day for 12 weeks, THEN one 14 mg nicotine patch per day for 2 weeks, THEN one 7 mg nicotine patch per day for 2 weeks.
  IF < or = 10 cigs/day: one 14 mg nicotine patch per day for 12 weeks, then one 7 mg for 4 weeks.
  Gum:
  IF > 24 cigs/day: ten 4 mg nicotine gum per day for 16 weeks. IF < or = 24 cigs/day: ten 2 mg nicotine patch per day for 16 weeks.
  Arms: 12, Patch, No Gum, Prequit, Int In-Person, Int Phone, 16Wk; 14, Patch, No Gum, No Prequit, Min In-Person, Int Phone, 16Wk; 15, Patch, No Gum, No Prequit, Int In-Person, Min Phone, 16Wk; 17, No Patch, Gum, Prequit, Min In-Person, Min Phone, 16Wk; 2, Patch, Gum, Prequit, Min In-Person, Int Phone, 16Wk; 20, No Patch, Gum, Prequit, Int In-Person, Int Phone, 16Wk; 22, No Patch, Gum, No Prequit, Min In-Person, Int Phone, 16Wk; 23, No Patch, Gum, No Prequit, Int In-Person, Min Phone, 16Wk; 26, No Patch, No Gum, Prequit, Min In-Person, Int Phone, 16Wk; 27, No Patch, No Gum, Prequit, Int In-Person, Min Phone, 16Wk; 29, No Patch, No Gum, No Prequit, Min In-Person, Min Phone, 16; 3, Patch, Gum, Prequit, Int In-Person, Min Phone, 16Wk; 32, No Patch, No Gum, No Prequit, Int In-Person, Int Phone, 16; 5, Patch, Gum, No Prequit, Min In-Person, Min Phone, 16Wk; 8, Patch, Gum, No Prequit, Int In-Person, Int Phone, 16Wk; 9, Patch, No Gum, Prequit, Min In-Person, Min Phone, 16Wk
Drug: Short Term Nicotine Patch + Nicotine Gum during the quit attempt — If randomized to this condition:
  After the target quit day:
  Patch:
  IF > 10 cigs/day: one 21 mg nicotine patch per day for 4 weeks, THEN one 14 mg nicotine patch per day for 2 weeks, THEN one 7 mg nicotine patch per day for 2 weeks.
  IF < or = 10 cigs/day: one 14 mg nicotine patch per day for 4 weeks, then one 7 mg for 4 weeks.
  Gum:
  IF > 24 cigs/day: ten 4 mg nicotine gum per day for 8 weeks. IF < or = 24 cigs/day: ten 2 mg nicotine gum per day for 8 weeks.
  Arms: 1, Patch, Gum, Prequit, Min In-Person, Min Phone, 8Wk; 10, Patch, No Gum, Prequit, Min In-Person, Int Phone, 8Wk; 11, Patch, No Gum, Prequit, Int In-Person, Min Phone, 8Wk; 13, Patch, No Gum, No Prequit, Min In-Person, Min Phone, 8Wk; 16, Patch, No Gum, No Prequit, Int In-Person, Int Phone, 8Wk; 18, No Patch, Gum, Prequit, Min In-Person, Int Phone, 8Wk; 19, No Patch, Gum, Prequit, Int In-Person, Min Phone, 8Wk; 21, No Patch, Gum, No Prequit, Min In-Person, Min Phone, 8Wk; 24, No Patch, Gum, No Prequit, Int In-Person, Int Phone, 8Wk; 25, No Patch, No Gum, Prequit, Min In-Person, Min Phone, 8Wk; 28, No Patch, No Gum, Prequit, Int In-Person, Int Phone, 8Wk; 30, No Patch, No Gum, No Prequit, Min In-Person, Int Phone, 8W; 31, No Patch, No Gum, No Prequit, Int In-Person, Min Phone, 8W; 4, Patch, Gum, Prequit, Int In-Person, Int Phone, 8Wk; 6, Patch, Gum, No Prequit, Min In-Person, Int Phone, 8Wk; 7, Patch, Gum, No Prequit, Int In-Person, Min Phone, 8Wk
Drug: Pre-Quit Nicotine Gum — If randomized to only the Pre-Quit Nicotine Gum condition (and not the Pre-Quit Nicotine Patch):
  Before quitting: Everyone will have ten 2 mg nicotine gum per day for 2 weeks before the target quit day.
  Arms: 17, No Patch, Gum, Prequit, Min In-Person, Min Phone, 16Wk; 18, No Patch, Gum, Prequit, Min In-Person, Int Phone, 8Wk; 19, No Patch, Gum, Prequit, Int In-Person, Min Phone, 8Wk; 20, No Patch, Gum, Prequit, Int In-Person, Int Phone, 16Wk; 21, No Patch, Gum, No Prequit, Min In-Person, Min Phone, 8Wk; 22, No Patch, Gum, No Prequit, Min In-Person, Int Phone, 16Wk; 23, No Patch, Gum, No Prequit, Int In-Person, Min Phone, 16Wk; 24, No Patch, Gum, No Prequit, Int In-Person, Int Phone, 8Wk
Drug: Pre-Quit Nicotine Patch — If randomized to only the Pre-Quit Nicotine Patch condition (and not the Pre-Quit Nicotine Gum):
  Before quitting: Everyone will have one 14 mg nicotine patch per day for 2 weeks before the target quit day.
  Arms: 10, Patch, No Gum, Prequit, Min In-Person, Int Phone, 8Wk; 11, Patch, No Gum, Prequit, Int In-Person, Min Phone, 8Wk; 12, Patch, No Gum, Prequit, Int In-Person, Int Phone, 16Wk; 13, Patch, No Gum, No Prequit, Min In-Person, Min Phone, 8Wk; 14, Patch, No Gum, No Prequit, Min In-Person, Int Phone, 16Wk; 15, Patch, No Gum, No Prequit, Int In-Person, Min Phone, 16Wk; 16, Patch, No Gum, No Prequit, Int In-Person, Int Phone, 8Wk; 9, Patch, No Gum, Prequit, Min In-Person, Min Phone, 16Wk
Drug: Pre-Quit Nicotine Patch + Pre-Quit Nicotine Gum — If randomized to both the Prequit Patch and Prequit Gum Conditions:
  Before quitting: Everyone will have ten 2 mg nicotine gum per day for 2 weeks and one 14 mg nicotine patch per day for 2 weeks before the target quit day.
  Arms: 1, Patch, Gum, Prequit, Min In-Person, Min Phone, 8Wk; 2, Patch, Gum, Prequit, Min In-Person, Int Phone, 16Wk; 3, Patch, Gum, Prequit, Int In-Person, Min Phone, 16Wk; 4, Patch, Gum, Prequit, Int In-Person, Int Phone, 8Wk; 5, Patch, Gum, No Prequit, Min In-Person, Min Phone, 16Wk; 6, Patch, Gum, No Prequit, Min In-Person, Int Phone, 8Wk; 7, Patch, Gum, No Prequit, Int In-Person, Min Phone, 8Wk; 8, Patch, Gum, No Prequit, Int In-Person, Int Phone, 16Wk

SUMMARY:
The goal of this research is to identify the best smoking cessation intervention components to be combined into a state-on-the-art, comprehensive smoking cessation intervention. This research examines the ability of different interventions, provided both prior to and after the quit attempt, to maximize the ability to initially quit and then stay quit. The investigators will be examining six different treatment interventions: pre-quit nicotine patch, pre-quit nicotine gum, pre-quit counseling, post-quit in-person counseling, post-quit phone counseling and duration of post-quit nicotine replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Report smoking at least 5 cigarettes per day for the previous 6 months;
* Able to read and write English;
* Agree to attend visits, to respond to coaching calls, and to respond to Interactive Voice Response (IVR) phone prompts;
* Plans to remain in the intervention catchment area for at least 12 months;
* Currently interested in quitting smoking (defined as would like to try to quit in the next 30 days).
* All women of childbearing potential will be required to agree to use an acceptable method of birth control to prevent pregnancy during the study.

Exclusion Criteria:

* Currently taking bupropion, Wellbutrin, chantix or varenicline (current use of NRT is not exclusionary if the participant agrees to use only study medication for the duration of the study);
* Study candidate is pregnant, trying to get pregnant, or nursing.
* A history of psychosis or bipolar disorder
* A history of skin or allergic reactions while using a nicotine patch.
* Had a heart attack, stroke, or abnormal electrocardiogram within the past 4 weeks.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2010-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan E Piper, PhD, Study Director — University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health; Timothy B Baker, PhD, Principal Investigator — University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health — http://www.ctri.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1, Patch, Gum, Prequit, Min In-Person, Min Phone, 8Wk | 2, Patch, Gum, Prequit, Min In-Person, Int Phone, 16Wk | 3, Patch, Gum, Prequit, Int In-Person, Min Phone, 16Wk | 4, Patch, Gum, Prequit, Int In-Person, Int Phone, 8Wk | 5, Patch, Gum, No Prequit, Min In-Person, Min Phone, 16Wk | 6, Patch, Gum, No Prequit, Min In-Person, Int Phone, 8Wk | 7, Patch, Gum, No Prequit, Int In-Person, Min Phone, 8Wk | 8, Patch, Gum, No Prequit, Int In-Person, Int Phone, 16Wk | 9, Patch, No Gum, Prequit, Min In-Person, Min Phone, 16Wk | 10, Patch, No Gum, Prequit, Min In-Person, Int Phone, 8Wk | 11, Patch, No Gum, Prequit, Int In-Person, Min Phone, 8Wk | 12, Patch, No Gum, Prequit, Int In-Person, Int Phone, 16Wk | 13, Patch, No Gum, No Prequit, Min In-Person, Min Phone, 8Wk | 14, Patch, No Gum, No Prequit, Min In-Person, Int Phone, 16Wk | 15, Patch, No Gum, No Prequit, Int In-Person, Min Phone, 16Wk | 16, Patch, No Gum, No Prequit, Int In-Person, Int Phone, 8Wk | 17, No Patch, Gum, Prequit, Min In-Person, Min Phone, 16Wk | 18, No Patch, Gum, Prequit, Min In-Person, Int Phone, 8Wk | 19, No Patch, Gum, Prequit, Int In-Person, Min Phone, 8Wk | 20, No Patch, Gum, Prequit, Int In-Person, Int Phone, 16Wk | 21, No Patch, Gum, No Prequit, Min In-Person, Min Phone, 8Wk | 22, No Patch, Gum, No Prequit, Min In-Person, Int Phone, 16Wk | 23, No Patch, Gum, No Prequit, Int In-Person, Min Phone, 16Wk | 24, No Patch, Gum, No Prequit, Int In-Person, Int Phone, 8Wk | 25, No Patch, No Gum, Prequit, Min In-Person, Min Phone, 8Wk | 26, No Patch, No Gum, Prequit, Min In-Person, Int Phone, 16Wk | 27, No Patch, No Gum, Prequit, Int In-Person, Min Phone, 16Wk | 28, No Patch, No Gum, Prequit, Int In-Person, Int Phone, 8Wk | 29, No Patch, No Gum, No Prequit, Min In-Person, Min Phone, 16 | 30, No Patch, No Gum, No Prequit, Min In-Person, Int Phone, 8W | 31, No Patch, No Gum, No Prequit, Int In-Person, Min Phone, 8W | 32, No Patch, No Gum, No Prequit, Int In-Person, Int Phone, 16
Started | 24 | 19 | 18 | 22 | 24 | 22 | 22 | 22 | 20 | 23 | 19 | 20 | 17 | 19 | 17 | 21 | 16 | 24 | 23 | 15 | 24 | 20 | 23 | 21 | 18 | 19 | 18 | 19 | 17 | 17 | 17 | 17
Completed | 22 | 16 | 16 | 20 | 20 | 20 | 20 | 20 | 19 | 19 | 18 | 20 | 16 | 16 | 17 | 15 | 13 | 19 | 20 | 13 | 22 | 18 | 19 | 19 | 15 | 19 | 14 | 18 | 17 | 17 | 16 | 14
Not Completed | 2 | 3 | 2 | 2 | 4 | 2 | 2 | 2 | 1 | 4 | 1 | 0 | 1 | 3 | 0 | 6 | 3 | 5 | 3 | 2 | 2 | 2 | 4 | 2 | 3 | 0 | 4 | 1 | 0 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1, Patch, Gum, Prequit, Min In-Person, Min Phone, 8Wk | 2, Patch, Gum, Prequit, Min In-Person, Int Phone, 16Wk | 3, Patch, Gum, Prequit, Int In-Person, Min Phone, 16Wk | 4, Patch, Gum, Prequit, Int In-Person, Int Phone, 8Wk | 5, Patch, Gum, No Prequit, Min In-Person, Min Phone, 16Wk | 6, Patch, Gum, No Prequit, Min In-Person, Int Phone, 8Wk | 7, Patch, Gum, No Prequit, Int In-Person, Min Phone, 8Wk | 8, Patch, Gum, No Prequit, Int In-Person, Int Phone, 16Wk | 9, Patch, No Gum, Prequit, Min In-Person, Min Phone, 16Wk | 10, Patch, No Gum, Prequit, Min In-Person, Int Phone, 8Wk | 11, Patch, No Gum, Prequit, Int In-Person, Min Phone, 8Wk | 12, Patch, No Gum, Prequit, Int In-Person, Int Phone, 16Wk | 13, Patch, No Gum, No Prequit, Min In-Person, Min Phone, 8Wk | 14, Patch, No Gum, No Prequit, Min In-Person, Int Phone, 16Wk | 15, Patch, No Gum, No Prequit, Int In-Person, Min Phone, 16Wk | 16, Patch, No Gum, No Prequit, Int In-Person, Int Phone, 8Wk | 17, No Patch, Gum, Prequit, Min In-Person, Min Phone, 16Wk | 18, No Patch, Gum, Prequit, Min In-Person, Int Phone, 8Wk | 19, No Patch, Gum, Prequit, Int In-Person, Min Phone, 8Wk | 20, No Patch, Gum, Prequit, Int In-Person, Int Phone, 16Wk | 21, No Patch, Gum, No Prequit, Min In-Person, Min Phone, 8Wk | 22, No Patch, Gum, No Prequit, Min In-Person, Int Phone, 16Wk | 23, No Patch, Gum, No Prequit, Int In-Person, Min Phone, 16Wk | 24, No Patch, Gum, No Prequit, Int In-Person, Int Phone, 8Wk | 25, No Patch, No Gum, Prequit, Min In-Person, Min Phone, 8Wk | 26, No Patch, No Gum, Prequit, Min In-Person, Int Phone, 16Wk | 27, No Patch, No Gum, Prequit, Int In-Person, Min Phone, 16Wk | 28, No Patch, No Gum, Prequit, Int In-Person, Int Phone, 8Wk | 29, No Patch, No Gum, No Prequit, Min In-Person, Min Phone, 16 | 30, No Patch, No Gum, No Prequit, Min In-Person, Int Phone, 8W | 31, No Patch, No Gum, No Prequit, Int In-Person, Min Phone, 8W | 32, No Patch, No Gum, No Prequit, Int In-Person, Int Phone, 16 | Total
Number analyzed (Participants) | 24 | 19 | 18 | 22 | 24 | 22 | 22 | 22 | 20 | 23 | 19 | 20 | 17 | 19 | 17 | 21 | 16 | 24 | 23 | 15 | 24 | 20 | 23 | 21 | 18 | 19 | 18 | 19 | 17 | 17 | 17 | 17 | 637
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Between 18 and 65 years | 24 | 19 | 18 | 20 | 22 | 22 | 22 | 22 | 17 | 22 | 18 | 19 | 16 | 19 | 17 | 20 | 15 | 23 | 22 | 15 | 23 | 20 | 21 | 20 | 18 | 19 | 14 | 17 | 15 | 15 | 16 | 17 | 607
  >=65 years | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 4 | 2 | 2 | 2 | 1 | 0 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.54 (9.90) | 44.79 (11.67) | 44.28 (10.88) | 43.91 (13.19) | 50.0 (12.03) | 41.50 (12.50) | 46.86 (11.67) | 39.73 (13.58) | 43.00 (14.18) | 47.43 (10.75) | 46.26 (11.84) | 45.10 (12.23) | 42.53 (12.58) | 42.63 (9.75) | 44.94 (10.97) | 50.05 (8.87) | 47.13 (10.68) | 45.83 (11.45) | 43.83 (13.66) | 45.20 (14.56) | 47.38 (9.57) | 46.30 (12.09) | 44.17 (12.51) | 45.33 (9.98) | 45.00 (11.78) | 46.32 (12.87) | 54.56 (11.59) | 48.37 (12.95) | 41.82 (15.02) | 48.29 (13.96) | 51.18 (10.00) | 40.65 (11.25) | 45.73 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 11 | 12 | 13 | 12 | 12 | 12 | 12 | 12 | 10 | 11 | 11 | 10 | 10 | 11 | 9 | 12 | 11 | 9 | 13 | 11 | 13 | 11 | 10 | 10 | 11 | 10 | 8 | 8 | 10 | 10 | 348
  Male | 12 | 8 | 7 | 10 | 11 | 10 | 10 | 10 | 8 | 11 | 9 | 9 | 6 | 9 | 7 | 10 | 7 | 12 | 12 | 6 | 11 | 9 | 10 | 10 | 8 | 9 | 7 | 9 | 9 | 9 | 7 | 7 | 289
Region of Enrollment [Number; unit: participants]
  United States | 24 | 19 | 18 | 22 | 24 | 22 | 22 | 22 | 20 | 23 | 19 | 20 | 17 | 19 | 17 | 21 | 16 | 24 | 23 | 15 | 24 | 20 | 23 | 21 | 18 | 19 | 18 | 19 | 17 | 17 | 17 | 17 | 637

OUTCOME MEASURES:

1. Secondary Outcome: Latency to Relapse
Description: Latency to Relapse during the first 6 months post-quit, with relapse defined as 7 consecutive days of smoking; this outcome will be analyzed in a Cox regression survival analysis model with non-relapsers coded as right-censored.
Time Frame: During the first 6 months post-quit
Measure: Number; unit: participants
Groups:
- No Pre-Quit Nicotine Patch: Participants randomized to this condition received No Pre-Quit Nicotine Patch; participants in this group received all combinations of the other five study treatments: No Pre-Quit Nicotine Gum or Pre-Quit Nicotine Gum; No Counseling Before the Quit Attempt or Counseling Before the Quit Attempt; Minimal In-person Counseling During the Quit Attempt or Intensive In-person Counseling During the Quit Attempt; Minimal Phone Counseling During the Quit Attempt or Intensive Phone Counseling During the Quit Attempt; Short Term or Long Term Nicotine Patch + Nicotine Gum During the Quit Attempt. The No Pre-Quit Nicotine Patch group consists of 308 participants (approximately half the total sample of 637) who will be compared with a group that received Pre-Quit Nicotine Patch (N=329; approximately half the total sample) in a main effect statistical comparison (No Pre-Quit Nicotine Patch vs. Pre-Quit Nicotine Patch).
- Pre-Quit Nicotine Patch: Participants randomized to this condition received Pre-Quit Nicotine Patch; participants in this group received all combinations of the other five study treatments: No Pre-Quit Nicotine Gum or Pre-Quit Nicotine Gum; No Counseling Before the Quit Attempt or Counseling Before the Quit Attempt; Minimal In-person Counseling During the Quit Attempt or Intensive In-person Counseling During the Quit Attempt; Minimal Phone Counseling During the Quit Attempt or Intensive Phone Counseling During the Quit Attempt; Short Term or Long Term Nicotine Patch + Nicotine Gum During the Quit Attempt. The Pre-Quit Nicotine Patch group consists of 329 participants (approximately half the total sample of 637) who will be compared with a group that received No Pre-Quit Nicotine Patch (N=308; approximately half the total sample) in a main effect statistical comparison (No Pre-Quit Nicotine Patch vs. Pre-Quit Nicotine Patch).
- No Pre-Quit Nicotine Gum: Participants randomized to this condition received No Pre-Quit Nicotine Gum; participants in this group received all combinations of the other five study treatments: No Pre-Quit Nicotine Patch or Pre-Quit Nicotine Patch; No Counseling Before the Quit Attempt or Counseling Before the Quit Attempt; Minimal In-person Counseling During the Quit Attempt or Intensive In-person Counseling During the Quit Attempt; Minimal Phone Counseling During the Quit Attempt or Intensive Phone Counseling During the Quit Attempt; Short Term or Long Term Nicotine Patch + Nicotine Gum During the Quit Attempt. The No Pre-Quit Nicotine Gum group consists of 298 participants (approximately half the total sample of 637) who will be compared with a group that received Pre-Quit Nicotine Gum (N=339; approximately half the total sample) in a main effect statistical comparison (No Pre-Quit Nicotine Gum vs. Pre-Quit Nicotine Gum).
- Pre-Quit Nicotine Gum: Participants randomized to this condition received Pre-Quit Nicotine Gum; participants in this group received all combinations of the other five study treatments: No Pre-Quit Nicotine Patch or Pre-Quit Nicotine Patch; No Counseling Before the Quit Attempt or Counseling Before the Quit Attempt; Minimal In-person Counseling During the Quit Attempt or Intensive In-person Counseling During the Quit Attempt; Minimal Phone Counseling During the Quit Attempt or Intensive Phone Counseling During the Quit Attempt; Short Term or Long Term Nicotine Patch + Nicotine Gum During the Quit Attempt. The Pre-Quit Nicotine Gum group consists of 339 participants (approximately half the total sample of 637) who will be compared with a group that received No Pre-Quit Nicotine Gum (N=298; approximately half the total sample) in a main effect statistical comparison (No Pre-Quit Nicotine Gum vs. Pre-Quit Nicotine Gum).
- No Counseling Before the Quit Attempt: Participants randomized to this condition received No Counseling Before the Quit Attempt; participants in this group received all combinations of the other five study treatments: No Pre-Quit Nicotine Patch or Pre-Quit Nicotine Patch; No Pre-Quit Nicotine Gum or Pre-Quit Nicotine Gum; Minimal In-person Counseling During the Quit Attempt or Intensive In-person Counseling During the Quit Attempt; Minimal Phone Counseling During the Quit Attempt or Intensive Phone Counseling During the Quit Attempt; Short Term or Long Term Nicotine Patch + Nicotine Gum During the Quit Attempt. The No Counseling Before the Quit Attempt group consists of 320 participants (approximately half the total sample of 637) who will be compared with a group that received Counseling Before the Quit Attempt (N=317; approximately half the total sample) in a main effect statistical comparison (No Counseling Before the Quit Attempt vs. Counseling Before the Quit Attempt).
- Counseling Before the Quit Attempt: Participants randomized to this condition received Counseling Before the Quit Attempt; participants in this group received all combinations of the other five study treatments: No Pre-Quit Nicotine Patch or Pre-Quit Nicotine Patch; No Pre-Quit Nicotine Gum or Pre-Quit Nicotine Gum; Minimal In-person Counseling During the Quit Attempt or Intensive In-person Counseling During the Quit Attempt; Minimal Phone Counseling During the Quit Attempt or Intensive Phone Counseling During the Quit Attempt; Short Term or Long Term Nicotine Patch + Nicotine Gum During the Quit Attempt. The Counseling Before the Quit Attempt group consists of 317 participants (approximately half the total sample of 637) who will be compared with a group that received No Counseling Before the Quit Attempt (N=320; approximately half the total sample) in a main effect statistical comparison (No Counseling Before the Quit Attempt vs. Counseling Before the Quit Attempt).
- Minimal In-person Counseling During the Quit Attempt: Participants randomized to this condition received Minimal In-person Counseling During the Quit Attempt; participants in this group received all combinations of the other 5 study treatments: No Pre-Quit Nicotine Patch or Pre-Quit Nicotine Patch; No Pre-Quit Nicotine Gum or Pre-Quit Nicotine Gum; No Counseling Before the Quit Attempt or Counseling Before the Quit Attempt; Minimal Phone Counseling During the Quit Attempt or Intensive Phone Counseling During the Quit Attempt; Short Term or Long Term Nicotine Patch + Nicotine Gum During the Quit Attempt. The Minimal In-person Counseling During the Quit Attempt group consists of 323 participants (approximately half the total sample of 637) who will be compared with a group that received Intensive In-person Counseling During the Quit Attempt(N=320; approximately half the total sample) in a main effect statistical comparison (Minimal In-person Counseling During the Quit Attempt vs Intensive In-person Counseling During the Quit Attempt).
- Intensive In-person Counseling During the Quit Attempt: Participants randomized to this condition received Intensive In-person Counseling During the Quit Attempt; participants in this group received all combinations of the other 5 study treatments: No Pre-Quit Nicotine Patch or Pre-Quit Nicotine Patch; No Pre-Quit Nicotine Gum or Pre-Quit Nicotine Gum; No Counseling Before the Quit Attempt or Counseling Before the Quit Attempt; Minimal Phone Counseling During the Quit Attempt or Intensive Phone Counseling During the Quit Attempt; Short Term or Long Term Nicotine Patch + Nicotine Gum During the Quit Attempt. The Intensive In-person Counseling During the Quit Attempt group consists of 314 participants (approximately half the total sample of 637) who will be compared with a group that received Minimal In-person Counseling During the Quit Attempt (N=323; approximately half the total sample) in a main effect statistical comparison (Minimal In-person Counseling During the Quit Attempt vs Intensive In-person Counseling During the Quit Attempt).
- Minimal Phone Counseling During the Quit Attemp: Participants randomized to this condition received Minimal Phone Counseling During the Quit Attempt; participants in this group received all combinations of the other five study treatments: No Pre-Quit Nicotine Patch or Pre-Quit Nicotine Patch; No Pre-Quit Nicotine Gum or Pre-Quit Nicotine Gum; No Counseling Before the Quit Attempt or Counseling Before the Quit Attempt; Minimal In-person Counseling During the Quit Attempt or Intensive In-person Counseling During the Quit Attempt; Short Term or Long Term Nicotine Patch + Nicotine Gum During the Quit Attempt. The Minimal Phone Counseling During the Quit Attempt group consists of 317 participants (approximately half the total sample of 637) who will be compared with a group that received Intensive Phone Counseling During the Quit Attempt (N=320; approximately half the total sample) in a main effect statistical comparison (Minimal Phone Counseling During the Quit Attempt vs Intensive Phone Counseling During the Quit Attempt).
- Intensive Phone Counseling During the Quit Attempt: Participants randomized to this condition received Intensive Phone Counseling During the Quit Attempt; participants in this group received all combinations of the other five study treatments: No Pre-Quit Nicotine Patch or Pre-Quit Nicotine Patch; No Pre-Quit Nicotine Gum or Pre-Quit Nicotine Gum; No Counseling Before the Quit Attempt or Counseling Before the Quit Attempt; Minimal In-person Counseling During the Quit Attempt or Intensive In-person Counseling During the Quit Attempt; Short Term or Long Term Nicotine Patch + Nicotine Gum During the Quit Attempt. The Intensive Phone Counseling During the Quit Attempt group consists of 320 participants (approximately half the total sample of 637) who will be compared with a group that received Minimal Phone Counseling During the Quit Attempt (N=317; approximately half the total sample) in a main effect statistical comparison (Minimal Phone Counseling During the Quit Attempt vs Intensive Phone Counseling During the Quit Attempt).
- Short Term (8 Weeks) Postquit Nicotine Patch + Nicotine Gum: Participants randomized to this condition received Short Term Nicotine Patch + Nicotine Gum (Combo NRT) During the Quit Attempt; participants in this group received all combinations of the other five study treatments: No Pre-Quit Nicotine Patch or Pre-Quit Nicotine Patch; No Pre-Quit Nicotine Gum or Pre-Quit Nicotine Gum; No Counseling Before the Quit Attempt or Counseling Before the Quit Attempt; Minimal In-person Counseling During the Quit Attempt or Intensive In-person Counseling During the Quit Attempt; Minimal Phone Counseling During the Quit Attempt or Intensive Phone Counseling During the Quit Attempt. The Short Term Combo NRT group consists of 333 participants (approximately half the total sample of 637) who will be compared with a group that received Long Term Combo NRT group (N=304; approximately half the total sample) in a main effect statistical comparison (Short Term Combo NRT vs. Long Term Combo NRT).
- Long Term (26 Weeks) Postquit Nicotine Patch + Nicotine Gum: Participants randomized to this condition received Long Term Nicotine Patch + Nicotine Gum (Combo NRT) During the Quit Attempt; participants in this group received all combinations of the other five study treatments: No Pre-Quit Nicotine Patch or Pre-Quit Nicotine Patch; No Pre-Quit Nicotine Gum or Pre-Quit Nicotine Gum; No Counseling Before the Quit Attempt or Counseling Before the Quit Attempt; Minimal In-person Counseling During the Quit Attempt or Intensive In-person Counseling During the Quit Attempt; Minimal Phone Counseling During the Quit Attempt or Intensive Phone Counseling During the Quit Attempt. The Long Term Combo NRT group consists of 304 participants (approximately half the total sample of 637) who will be compared with a group that received Long Term Combo NRT group (N=333; approximately half the total sample) in a main effect statistical comparison (Short Term Combo NRT vs. Long Term Combo NRT).
Arm/Group | No Pre-Quit Nicotine Patch | Pre-Quit Nicotine Patch | No Pre-Quit Nicotine Gum | Pre-Quit Nicotine Gum | No Counseling Before the Quit Attempt | Counseling Before the Quit Attempt | Minimal In-person Counseling During the Quit Attempt | Intensive In-person Counseling During the Quit Attempt | Minimal Phone Counseling During the Quit Attemp | Intensive Phone Counseling During the Quit Attempt | Short Term (8 Weeks) Postquit Nicotine Patch + Nicotine Gum | Long Term (26 Weeks) Postquit Nicotine Patch + Nicotine Gum
Number analyzed (Participants) | 308 | 329 | 298 | 339 | 320 | 317 | 323 | 314 | 317 | 320 | 333 | 304
participants
  # Participants Who Relapsed (Smoking) | 235 | 243 | 228 | 250 | 243 | 235 | 246 | 232 | 242 | 236 | 246 | 232
  # Participants Who Did Not Relapse (Not Smoking) | 73 | 86 | 70 | 89 | 77 | 82 | 77 | 82 | 75 | 84 | 87 | 72
Statistical Analysis 1: Comparison: No Pre-Quit Nicotine Patch vs Pre-Quit Nicotine Patch; The Cox regression model effects consisted of six treatment effects, 15 two-way treatment interactions, and three covariates : gender and two items from the Fagerstrom Test of Nicotine Dependence (Item 1: time to first cigarette; Item 4: cigarettes per day); Test type: Superiority or Other; p = .312, Regression, Cox; Cox Proportional Hazard = .954, 95% CI 2-sided [.871 to 1.045]
Statistical Analysis 2: Comparison: No Pre-Quit Nicotine Gum vs Pre-Quit Nicotine Gum; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .664, Regression, Cox; Cox Proportional Hazard = .980, 95% CI 2-sided [.894 to 1.074]
Statistical Analysis 3: Comparison: No Counseling Before the Quit Attempt vs Counseling Before the Quit Attempt; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .814, Regression, Cox; Cox Proportional Hazard = .989, 95% CI 2-sided [.903 to 1.084]
Statistical Analysis 4: Comparison: Minimal In-person Counseling During the Quit Attempt vs Intensive In-person Counseling During the Quit Attempt; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .093, Regression, Cox; Cox Proportional Hazard = .925, 95% CI 2-sided [.844 to 1.013]
Statistical Analysis 5: Comparison: Minimal Phone Counseling During the Quit Attemp vs Intensive Phone Counseling During the Quit Attempt; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .716, Regression, Cox; Cox Proportional Hazard = .983, 95% CI 2-sided [.898 to 1.077]
Statistical Analysis 6: Comparison: Short Term (8 Weeks) Postquit Nicotine Patch + Nicotine Gum vs Long Term (26 Weeks) Postquit Nicotine Patch + Nicotine Gum; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .511, Regression, Cox; Cox Proportional Hazard = 1.031, 95% CI 2-sided [.941 to 1.130]

2. Primary Outcome: Self-Reported 7-Day Point-Prevalence Abstinence
Description: Self-Reported 7-Day Point-Prevalence Abstinence is a dichotomous outcome with values of 0 and 1 where 0=smoking on one or more of the past 7 days at the assessment endpoint (16 weeks post-quit) and 1=no smoking on any of the past 7 days at the assessment endpoint (i.e., abstinent for the past 7 days); this outcome will be analyzed in a logistic regression analysis model.
  Note: This abstinence primary outcome replaces latency to relapse (now designated as a secondary outcome) because reviewers of the now-accepted manuscript (at the journal "Addiction") advised us to change the primary outcome to the current week 16 Self-Reported 7-Day Point-Prevalence Abstinence outcome.
Time Frame: 16 weeks post-quit
Measure: Number; unit: participants
Arm/Group | No Pre-Quit Nicotine Patch | Pre-Quit Nicotine Patch | No Pre-Quit Nicotine Gum | Pre-Quit Nicotine Gum | No Counseling Before the Quit Attempt | Counseling Before the Quit Attempt | Minimal In-person Counseling During the Quit Attempt | Intensive In-person Counseling During the Quit Attempt | Minimal Phone Counseling During the Quit Attemp | Intensive Phone Counseling During the Quit Attempt | Short Term (8 Weeks) Postquit Nicotine Patch + Nicotine Gum | Long Term (26 Weeks) Postquit Nicotine Patch + Nicotine Gum
Number analyzed (Participants) | 308 | 329 | 298 | 339 | 320 | 317 | 323 | 314 | 317 | 320 | 333 | 304
participants
  # Participants Who Were Smoking | 208 | 209 | 201 | 216 | 221 | 196 | 217 | 200 | 211 | 206 | 223 | 194
  # Participants Who Were Abstinent | 100 | 120 | 97 | 123 | 99 | 121 | 106 | 114 | 106 | 114 | 110 | 110
Statistical Analysis 1: Comparison: No Pre-Quit Nicotine Patch vs Pre-Quit Nicotine Patch; The logistic regression model effects consisted of six treatment main effects and 15 two-way treatment interactions. The main effects provide direct tests of the primary aim of the study, i.e., determining whether or not more intensive treatments (compared to less intensive treatments; e.g., No Pre-Quit Nicotine Patch vs. Pre-Quit Nicotine Patch) would result in significantly higher abstinence at 16 weeks post-quit; Test type: Superiority or Other; p = .341, Regression, Logistic; Odds Ratio (OR) = 1.087, 95% CI 2-sided [.916 to 1.290]
Statistical Analysis 2: Comparison: No Pre-Quit Nicotine Gum vs Pre-Quit Nicotine Gum; The logistic regression model effects consisted of six treatment main effects and 15 two-way treatment interactions. The main effects provide direct tests of the primary aim of the study, i.e., determining whether or not more intensive treatments (compared to less intensive treatments; e.g., No Pre-Quit Nicotine Gum vs. Pre-Quit Nicotine Gum) would result in significantly higher abstinence at 16 weeks post-quit; Test type: Superiority or Other; p = .207, Regression, Logistic; Odds Ratio (OR) = 1.117, 95% CI 2-sided [.941 to 1.325]
Statistical Analysis 3: Comparison: No Counseling Before the Quit Attempt vs Counseling Before the Quit Attempt; The logistic regression model effects consisted of six treatment main effects and 15 two-way treatment interactions. The main effects provide direct tests of the primary aim of the study, i.e., determining whether or not more intensive treatments (compared to less intensive treatments; e.g., No Counseling Before the Quit Attempt vs. Counseling Before the Quit Attempt) would result in significantly higher abstinence at 16 weeks post-quit; Test type: Superiority or Other; p = .041, Regression, Logistic; Odds Ratio (OR) = 1.196, 95% CI 2-sided [1.008 to 1.420]
Statistical Analysis 4: Comparison: Minimal In-person Counseling During the Quit Attempt vs Intensive In-person Counseling During the Quit Attempt; The logistic regression model effects consisted of six treatment main effects and 15 two-way treatment interactions. The main effects provide direct tests of the primary aim of the study, i.e., determining whether or not more intensive treatments (compared to less intensive treatments; e.g., Minimal In-person Counseling During the Quit Attempt vs. Intensive In-person Counseling During the Quit Attempt) would result in significantly higher abstinence at 16 weeks post-quit; Test type: Superiority or Other; p = .536, Regression, Logistic; Odds Ratio (OR) = 1.056, 95% CI 2-sided [.889 to 1.254]
Statistical Analysis 5: Comparison: Minimal Phone Counseling During the Quit Attemp vs Intensive Phone Counseling During the Quit Attempt; The logistic regression model effects consisted of six treatment main effects and 15 two-way treatment interactions. The main effects provide direct tests of the primary aim of the study, i.e., determining whether or not more intensive treatments (compared to less intensive treatments; e.g., Minimal Phone Counseling During the Quit Attempt vs. Intensive Phone Counseling During the Quit Attempt) would result in significantly higher abstinence at 16 weeks post-quit; Test type: Superiority or Other; p = .587, Regression, Logistic; Odds Ratio (OR) = 1.049, 95% CI 2-sided [.883 to 1.246]
Statistical Analysis 6: Comparison: Short Term (8 Weeks) Postquit Nicotine Patch + Nicotine Gum vs Long Term (26 Weeks) Postquit Nicotine Patch + Nicotine Gum; The logistic regression model effects consisted of six treatment main effects and 15 two-way treatment interactions. The main effects provide direct tests of the primary aim of the study, i.e., determining whether or not more intensive treatments (compared to less intensive treatments; e.g., Short Term (8 Weeks) Postquit Nicotine Patch + Nicotine Gum vs. Long Term (26 Weeks) Postquit Nicotine Patch + Nicotine Gum) would result in significantly higher abstinence at 16 weeks post-quit; Test type: Superiority or Other; p = .389, Regression, Logistic; Odds Ratio (OR) = 1.078, 95% CI 2-sided [.909 to 1.278]

ADVERSE EVENTS:
Time Frame: AEs were reported for the duration of time when the participant was on medication, 1 week before the quit attempt (if given prequit meds) and 4 weeks after the quit attempt, for up to 16 weeks after the quit attempt.
Description: Protocol prompted AE assessments occurred at week 1 (if given prequit meds) and weeks 1 and 4 postquit. Data from ad Hoc AE reports and protocol prompted AE assessments were combined. Only AEs where 5% or more of those from a study arm were reported and compared to other study arms.
Groups:
- Pre-Quit Nicotine Gum and Pre-Quit Nicotine Patch: Pre-Quit Nicotine Gum and Pre-Quit Nicotine Patch
  Participants randomized to this condition received Pre-Quit Nicotine Gum and Pre-Quit Nicotine Patch.
  Before quitting: Everyone had ten 2 mg nicotine gum per day for 2 weeks and one 14 mg nicotine patch per day for 2 weeks before the target quit day.
- Pre-Quit Nicotine Patch: Pre-Quit Nicotine Patch
  Participants randomized to this condition received Pre-Quit Nicotine Patch.
  Before quitting: Everyone had one 14 mg nicotine patch per day for 2 weeks before the target quit day.
- Pre-Quit Nicotine Gum: Pre-Quit Nicotine Gum
  Participants randomized to this condition received Pre-Quit Nicotine Gum.
  Before quitting: Everyone had one 14 mg nicotine patch per day for 2 weeks before the target quit day.
- No Pre-Quit Nicotine Patch Nor Gum: No Pre-Quit Nicotine Patch nor Gum
  Participants randomized to this condition received neither the Pre-Quit Nicotine Patch nor the Pre-Quit Nicotine Gum.
- Long Term (16 Weeks) Postquit Nicotine Patch + Nicotine Gum: Long Term (16 Weeks) Postquit Nicotine Patch + Nicotine Gum
  Participants randomized to this condition received Long Term Nicotine Patch + Nicotine Gum (Combo NRT) During the Quit Attempt.
- Short Term (8 Weeks) Postquit Nicotine Patch + Nicotine Gum: Short Term (8 Weeks) Postquit Nicotine Patch + Nicotine Gum
  Participants randomized to this condition received Short Term Nicotine Patch + Nicotine Gum (Combo NRT) During the Quit Attempt.
Arm/Group | Pre-Quit Nicotine Gum and Pre-Quit Nicotine Patch | Pre-Quit Nicotine Patch | Pre-Quit Nicotine Gum | No Pre-Quit Nicotine Patch Nor Gum | Long Term (16 Weeks) Postquit Nicotine Patch + Nicotine Gum | Short Term (8 Weeks) Postquit Nicotine Patch + Nicotine Gum
Serious Adverse Events (participants affected / at risk) | 1/173 | 1/156 | 0/166 | 0/142 | 5/333 | 2/304
Other Adverse Events (participants affected / at risk) | 32/173 | 27/156 | 22/166 | 0/142 | 51/304 | 55/333
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-Quit Nicotine Gum and Pre-Quit Nicotine Patch (N=173) | Pre-Quit Nicotine Patch (N=156) | Pre-Quit Nicotine Gum (N=166) | No Pre-Quit Nicotine Patch Nor Gum (N=142) | Long Term (16 Weeks) Postquit Nicotine Patch + Nicotine Gum (N=333) | Short Term (8 Weeks) Postquit Nicotine Patch + Nicotine Gum (N=304)
Death- Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurological (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Quit Nicotine Gum and Pre-Quit Nicotine Patch (N=173) | Pre-Quit Nicotine Patch (N=156) | Pre-Quit Nicotine Gum (N=166) | No Pre-Quit Nicotine Patch Nor Gum (N=142) | Long Term (16 Weeks) Postquit Nicotine Patch + Nicotine Gum (N=304) | Short Term (8 Weeks) Postquit Nicotine Patch + Nicotine Gum (N=333)
Indigestion (Gastrointestinal disorders) | 4 | 1 | 10 | 0 | 8 | 5
Nausea (Gastrointestinal disorders) | 13 | 8 | 12 | 0 | 15 | 20
Skin Rash (Skin and subcutaneous tissue disorders) | 6 | 11 | 1 | 0 | 23 | 26
Vivid Dreams (Nervous system disorders) | 17 | 11 | 2 | 0 | 19 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes